CLINICAL TRIAL: NCT04861233
Title: Post-Marketing Surveillance (Usage Results Study) of Adult Patients Treated With Lubiprostone for Indications Approved in South Korea
Brief Title: A Study of Lubiprostone to Treat Constipation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JL-PMS-AM
Record Dates: First submitted 2021-04-26; First posted 2021-04-27 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Constipation
Keywords: Drug Therapy
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants diagnosed with constipation who have been prescribed with lubiprostone for the first time in a real-world setting will be observed prospectively and followed up for 12 months after initiation of study medication. Treatment regimen, frequency of laboratory and clinical assessments will be determined by investigator in a routine clinical practice.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The main aim of this study is to check the side effects from lubiprostone in adults with constipation. Participants will be treated with lubiprostone according to their clinic's standard practice.

DETAILED DESCRIPTION:
This is a prospective, observational post-marketing surveillance study of lubiprostone in participants with constipation. The study will assess the safety and effectiveness of lubiprostone for its approved indication with real-world setting in South Korea.

The study will enroll approximately 3000 participants. The data will be collected prospectively at the study sites will be recorded into electronic case report forms (e-CRFs). All the participants will be assigned to a single observational cohort:

• All Participants

The study will be conducted in South Korea. The overall duration of the study will be approximately 6 years. Data collection will be based on routinely scheduled visits during a 12-month follow up period for each participant up to a final follow-up when the participant discontinues treatment or at the end of follow-up period for any participants still taking lubiprostone.

NOTE: This product was divested from Takeda to Jeil in 2022.

ELIGIBILITY:
Inclusion Criteria:

1. South Korean adult.
2. With constipation caused by:

   * Chronic Idiopathic Constipation (CIC), or
   * Opioid-Induced Constipation (OIC) from treatment for chronic, non-cancer pain, including participants with chronic pain related to prior cancer or its treatment who do not require frequent (example weekly) opioid dosage escalation.
3. Is newly prescribed (first incident) and initiates lubiprostone for the treatment of constipation.

Exclusion Criteria:

1. Treated with lubiprostone outside of the locally approved label in South Korea.
2. Participating in any other clinical study investigating one (or more) of the approved indications of lubiprostone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants with first incident prescription for treatment with lubiprostone will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting One or More Adverse Events (AEs) | Up to 12 months
  AEs is defined as any undesirable and unintended signs (example, abnormal laboratory values), symptoms, or diseases which occur during or following the administration of the drug, this does not necessarily require causal relationship.
Number of Participants Reporting One or More Serious Adverse Events (SAEs) | Up to 12 months
  A SAE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.

SECONDARY OUTCOMES:
Change From Baseline in the Frequency of Spontaneous Bowel Movement (SBM) at End of Treatment | Baseline up to end of treatment (approximately 12 months)
  SBM is a bowel movement occurring in the absence of laxative use. Change from baseline values will be reported for participants who discontinue lubiprostone during study period.
Time to Resolution of Symptoms After Treatment Discontinuation | Up to 12 months
  Time to resolution of symptoms defined as discontinuation of treatment with lubiprostone.
Change From Baseline in Frequency of SBM After 12-month Follow up | Up to 12 months
  SBM is a bowel movement occurring in the absence of laxative use. Change from baseline values after 12-months follow up period will be reported for participants.

CONTACTS AND LOCATIONS:
Overall Officials: Site Contact, Study Director — Jeil Pharmaceutical Co., Ltd.
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/608c06ad688ad8001f42fbc0